CLINICAL TRIAL: NCT04574440
Title: Evaluation of Cerebral Oxygenation Using Functional Near Infrared Spectroscopy in Adult Surgery
Brief Title: Functional Near Infrared Spectroscopy in Adult Surgery
Status: Recruiting | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: FNIRS
Record Dates: First submitted 2020-02-27; First posted 2020-10-05 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Cerebral Injury
Keywords: multichannel functional near infrared spectroscopy (fNIRS); cerebral oxygenation; cardiac surgery
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- multichannel fNIRS monitoring: Patients who will be enrolled in this study will be monitored during cardiac surgery using multichannel fNIRS monitoring. This consists of wearing the NIRS cap during surgery. The patient's surgery and subsequent medical care will not be altered.
  Interventions: Device: multichannel fNIRS monitoring

INTERVENTIONS:
Device: multichannel fNIRS monitoring — Patients who will be enrolled in this study will be monitored during cardiac surgery using multichannel fNIRS monitoring. This consists of wearing the NIRS cap that will be positioned on the patient's head according to international operational guidelines and will be secured to the temporal region of the patient's forehead. The NIRS cap is entirely non-invasive and does not pose any additional risk to the patient. Monitoring will be commenced prior to the induction of anesthesia. Subsequent surgical and medical care will not be affected.

SUMMARY:
Brain injury is a serious problem after cardiac surgery. Brain injury can become evident in the form of stroke and cognitive dysfunction after surgery. The current neuromonitoring technique used is unable to monitor the region of the brain that is most susceptible to injury. This study aims to use a novel, non-invasive brain monitoring technique known as multichannel functional near infrared spectroscopy to assess brain oxygenation at multiple brain regions simultaneously during cardiac surgery. This research enables the investigators to understand the differences between regional brain oxygenation during cardiac surgery and to assess the feasibility and effectiveness of multichannel functional near infrared spectroscopy to be used as a future brain monitoring technique to detect brain injury in cardiac surgery.

DETAILED DESCRIPTION:
Perioperative cerebral injury is a common and significant complication of patients undergoing cardiac surgery. 1,2 During cardiac surgery, cerebral injury can occur as a result of hypoperfusion, cerebral embolism, and/or inflammation. 3 These intraoperative cerebral injuries could manifest as postoperative neurocognitive dysfunction (e.g., impaired memory and attention, mood alterations), stroke, delirium, visual field deficits and coma. 4 Around 1% to 4% of cardiac surgical patients with closed-chamber cardiac procedures are complicated with stroke. The incidence of stroke increases markedly to about 8% to 9% in open-chamber (e.g., valvular surgery) or combined/complex procedures. These patients with neurological injury are associated with increased postoperative mortality, prolonged intensive care unit, hospital stay, decreased quality of life, and decreased long-term survival. 4 Despite the advancement of surgical techniques and perioperative care leading to a progressive decrease in cardiac surgical mortality since the 1980s1,5,6, the incidence of postoperative neurologic complications has remained relatively unchanged. This is largely related to the lack of effective monitoring and intervention to detect and mitigate intraoperative cerebral injury.

One potentially treatable cause of cerebral injury during cardiac surgery is hypoperfusion related infarct/ischemia. 7 Watershed, or boundary zone, are situated along border zones between the territories of two major cerebral arteries (e.g., the middle and posterior, or the anterior and middle cerebral arteries) where terminal arteriolar anastomoses exist which are more susceptible to hypoperfusion related infarct/ischemia. 8 These hypoperfusion related injuries are potentially treatable by increasing systematic blood pressure if those injuries are being identified early. Previous study has used electroencephalography to detect intraoperative brain injury at the watershed area9, but the clinical utility of electroencephalography is limited because of its cumbersome set-up and complex logistics. As such, this study aims to use a novel multichannel fNIRS to detect and monitor cerebral oxygenation at multiple brain regions simultaneously for adult patients undergoing during cardiac surgery. This study will increase the experiences of using fNIRS as a monitoring tool in cardiac surgery and improve the understandings to the cerebral injury pattern during cardiac surgery.

Multichannel functional near infrared spectroscopy (fNIRS) is an emerging brain-imaging technique to measure hemodynamic changes at the cortical surface. During the acquisition of fNIRS data light (600-900 nm) is emitted from light sources that can pass through the skull and reach cortex. Photons reflected from the cortex can be detected and quantified by detectors placed in close proximity to the sources. Light is mainly absorbed by oxygenated hemoglobin and deoxygenated hemoglobin, which have distinct absorption spectra. Alterations in the concentrations of oxy- and deoxy-hemoglobin derived from neuronal activation can be quantified using two or more wavelengths. The early studies has showed that the use of two channels cerebral near-infrared spectroscopy can avoid profound cerebral desaturation and is associated with significantly fewer incidences of major organ dysfunction. 10 However, one major limitation of two channels NIRS is that sensor placement is currently limited to forehead that only the frontal lobes are being monitored. Such placement prevents monitoring the critical posterior watershed at the juncture of the anterior, middle, and posterior cerebral arteries, and results in undetected stroke despite the patients having normal cerebral oxygenation throughout the surgery. The lack of comprehensive cortical coverage of the important brain regions such as water-shed area also limit the utility of two channels NIRS as a research tool to assess regional cerebral flow and metabolism during cardiac surgery. The multichannel fNIRS offers a number of advantages for assessing surgical patients intraoperatively including its high temporal resolution (~100ms), low-cost and portability. The multichannel fNIRS allows up to 64 channels of real-time data acquisition and interpretation, which allows adequate spatial and temporal resolutions to assess the brain regions at risk intraoperatively. In this study, only 16 channels will be used to assess the brain oxygenation.

The fNIRS system in this study is a class I Health Canada approved device (NIRx NIRScout 64x32 Laser/LED 4-wavelength fNRIS system, info:https://nirx.net/nirscout). It does not heat up nor can it damage eyesight. This commercially available device has been used safely in previous studies in neonatal population at Western (WREM #: 111168, 113443) and other studies published in the literature. This device is approved for brain oxygenation monitoring in humans.

Single site, prospective, observational study where patients undergoing cardiac surgical procedures will be monitored using multichannel fNIRS monitoring to assess cerebral oxygenation in regions of the brain that are susceptible to injury during cardiac surgery. No intervention will be used in this study. 40 patients total will be included in the study and receive this monitoring during surgery. There will be no randomization and no additional changes to standard of care.

Patients who agree to participate in this study will receive brain monitoring in the form of multichannel fNIRS monitoring that is not standard of care. This consists of wearing the NIRS cap that will be positioned on the patient's head according to international operational guidelines and will be secured to the temporal region of the patient's forehead. The NIRS cap is entirely non-invasive and does not pose any additional risk to the patient. Monitoring will be commenced prior to the induction of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Adult cardiac surgery patients who are scheduled to have elective cardiac operations.

Exclusion Criteria:

* Under 18 years of age
* have skin lesions or other conditions that preclude the application of fNIRS to the head
* lack of written consent
* emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cardiac surgery patients who are scheduled to have elective cardiac operations. The type of cardiac surgery is not restricted.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-12-20 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
feasibility of using multichannel fNIRS to detect and monitor cerebral oxygenation of multiple brain regions during cardiac surgery measured by detecting cortical hemodynamic and metabolic changes in different brain regions. | During the procedure/surgery
  Assess the feasibility of using multichannel fNIRS to detect and monitor cerebral oxygenation of multiple brain regions during cardiac surgery. This will be measured by using the multichannel fNIRS monitor during cardiac surgery and to determine if this monitor can detect cortical hemodynamic and metabolic changes in different brain regions. Data will be acquired using the NIRStar Software v14.0 (NIRx Medical Technologies LLC, Berlin, Germany) at a sampling rate of 10Hz.
Describe the regional cerebral oxygenation changes during cardiac surgery measured by using using multichannel fNIRS | During the procedure/surgery
  Describe the regional cerebral oxygenation changes during cardiac surgery. This will be measured by using multichannel fNIRS during cardiac surgery and determining whether it can detect differences in brain oxygenation in different regions of the brain. Data will be acquired using the NIRStar Software v14.0 (NIRx Medical Technologies LLC, Berlin, Germany) at a sampling rate of 10Hz .

CONTACTS AND LOCATIONS:
Overall Officials: Jason Chui, MD, Principal Investigator — Western University
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McKhann GM, Grega MA, Borowicz LM Jr, Baumgartner WA, Selnes OA. Stroke and encephalopathy after cardiac surgery: an update. Stroke. 2006 Feb;37(2):562-71. doi: 10.1161/01.STR.0000199032.78782.6c. Epub 2005 Dec 22. PMID 16373636
- [Background] Roach GW, Kanchuger M, Mangano CM, Newman M, Nussmeier N, Wolman R, Aggarwal A, Marschall K, Graham SH, Ley C. Adverse cerebral outcomes after coronary bypass surgery. Multicenter Study of Perioperative Ischemia Research Group and the Ischemia Research and Education Foundation Investigators. N Engl J Med. 1996 Dec 19;335(25):1857-63. doi: 10.1056/NEJM199612193352501. PMID 8948560
- [Background] Rankin JM, Silbert PL, Yadava OP, Hankey GJ, Stewart-Wynne EG. Mechanism of stroke complicating cardiopulmonary bypass surgery. Aust N Z J Med. 1994 Apr;24(2):154-60. doi: 10.1111/j.1445-5994.1994.tb00551.x. PMID 8042943
- [Background] Salazar JD, Wityk RJ, Grega MA, Borowicz LM, Doty JR, Petrofski JA, Baumgartner WA. Stroke after cardiac surgery: short- and long-term outcomes. Ann Thorac Surg. 2001 Oct;72(4):1195-201; discussion 1201-2. doi: 10.1016/s0003-4975(01)02929-0. PMID 11603436
- [Background] Tufo HM, Ostfeld AM, Shekelle R. Central nervous system dysfunction following open-heart surgery. JAMA. 1970 May 25;212(8):1333-40. No abstract available. PMID 5467674
- [Background] Gardner TJ, Horneffer PJ, Manolio TA, Pearson TA, Gott VL, Baumgartner WA, Borkon AM, Watkins L Jr, Reitz BA. Stroke following coronary artery bypass grafting: a ten-year study. Ann Thorac Surg. 1985 Dec;40(6):574-81. doi: 10.1016/s0003-4975(10)60352-9. PMID 3878134
- [Background] Sun LY, Chung AM, Farkouh ME, van Diepen S, Weinberger J, Bourke M, Ruel M. Defining an Intraoperative Hypotension Threshold in Association with Stroke in Cardiac Surgery. Anesthesiology. 2018 Sep;129(3):440-447. doi: 10.1097/ALN.0000000000002298. PMID 29889106
- [Background] Gottesman RF, Sherman PM, Grega MA, Yousem DM, Borowicz LM Jr, Selnes OA, Baumgartner WA, McKhann GM. Watershed strokes after cardiac surgery: diagnosis, etiology, and outcome. Stroke. 2006 Sep;37(9):2306-11. doi: 10.1161/01.STR.0000236024.68020.3a. Epub 2006 Jul 20. PMID 16857947
- [Background] Malone M, Prior P, Scholtz CL. Brain damage after cardiopulmonary by-pass: correlations between neurophysiological and neuropathological findings. J Neurol Neurosurg Psychiatry. 1981 Oct;44(10):924-31. doi: 10.1136/jnnp.44.10.924. PMID 7310410
- [Background] Murkin JM, Adams SJ, Novick RJ, Quantz M, Bainbridge D, Iglesias I, Cleland A, Schaefer B, Irwin B, Fox S. Monitoring brain oxygen saturation during coronary bypass surgery: a randomized, prospective study. Anesth Analg. 2007 Jan;104(1):51-8. doi: 10.1213/01.ane.0000246814.29362.f4. PMID 17179242